CLINICAL TRIAL: NCT02339168
Title: Enzalutamide and Metformin Combination Therapy to Overcome Autophagy Resistance in Castration Resistant Prostate Cancer
Brief Title: Enzalutamide and Metformin Hydrochloride in Treating Patients With Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Medivation, Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 680462; UCDCC#243 (Other: UC Davis UCDCC#243); UCDCC#243 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2014-02668 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- enzalutamide and metformin hydrochloride (Experimental): Patients receive enzalutamide PO QD and metformin hydrochloride PO BID. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: MDV3100; Xtandi
Drug: Metformin Hydrochloride — Given PO
  Other Names: Glucophage; Metformin HCl

SUMMARY:
This phase I trial studies the side effects and best dose of metformin hydrochloride when given together with enzalutamide in treating patients with prostate cancer that has not responded to previous treatment with hormones. Hormone therapy using enzalutamide may fight prostate cancer by lowering the amount of androgens the body makes and blocking the use of androgens by the tumor cells. Metformin hydrochloride, used for diabetes, may also help kill tumor cells. Giving enzalutamide together with metformin hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of enzalutamide when given in combination with metformin (metformin hydrochloride) to patients with castration resistant prostate cancer (CRPC), where fewer than 33% of patients experienced dose limiting toxicity (DLT) attributable to the study regimen and to recommend a phase II dose for the combination.

SECONDARY OBJECTIVES:

I. To determine prostate-specific antigen (PSA) response in patients with CRPC with given enzalutamide in combination with metformin.

II. To determine PSA progression in patients with CRPC with given enzalutamide in combination with metformin.

III. To investigate the feasibility and safety of enzalutamide when given in combination with metformin hydrochloride to patients with CRPC.

IV. To obtain preliminary evidence of efficacy for this combination.

TERTIARY OBJECTIVES:

I. To collect computed tomography (CT)-guided biopsies of metastatic soft tissue or bone tumor tissue for analysis of androgen receptor (AR) gene signature as an integrated biomarker (University of California San Francisco [UCSF] to conduct analysis).

II. To collect serum samples for the measurement of PSA levels and bone re-absorption markers.

OUTLINE: This is a dose-escalation study of metformin hydrochloride.

Patients receive enzalutamide orally (PO) once daily (QD) and metformin hydrochloride PO twice daily (BID). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed prostate cancer with a Gleason score available or interpretable; patients must have prostate cancer deemed to be castration-resistant by one or more of the following criteria (despite androgen deprivation and anti-androgen withdrawal when applicable):

  * Progression of unidimensionally measurable disease assessed within 28 days prior to initial administration of drug
  * Progression of evaluable but not measurable disease assessed within 28 days prior to initial administration of drug for PSA evaluation and within 42 days for imaging studies (e.g, bone scans)
  * NOTE: rising PSA, defined as at least two consecutive rises in PSA to be documented over a reference value (measure 1); the first rising PSA (measure 2) should be taken at least 7 days after the reference value; a third confirmatory PSA measure (2nd beyond the reference level) should be greater than the second measure, and it must be obtained at least 7 days after the 2nd measure; if this is not the case, a fourth PSA is required to be taken and be greater than the second measure; measurable disease is not required
* Patients who have measurable disease must have had X-rays, scans or physical examinations used for tumor measurement completed within 28 days prior to initial administration of drug
* Patients must have non-measurable disease (such as nuclear medicine bone scans) and non-target lesions (such as PSA level) assessed within 28 days prior to initial administration of drug
* Soft tissue disease that has been radiated within the two months prior to registration is not assessable as measurable disease; soft tissue disease that has been radiated two or more months prior to registration is assessable as measurable disease provided that the lesion has progressed following radiation; patients must have at least one measurable lesion outside the previously irradiated region in order to be considered to have measurable disease
* Patients must have been surgically or medically castrated; if the method of castration was luteinizing hormone-releasing hormone (LHRH) agonists (leuprolide or goserelin), then the patient must be willing to continue the use of LHRH agonists; serum testosterone must be at castrate levels (< 50 ng/dL) at least 14 days prior to registration
* If the patient has been treated with non-steroidal anti-androgens (flutamide, bicalutamide or nilutamide) or other hormonal treatment (such as ketoconazole), these agents must have been stopped at least 28 days prior to enrollment for flutamide or ketoconazole, and at least 42 days prior to enrollment for bicalutamide or nilutamide; and the patients must have demonstrated progression of disease since the agents were suspended
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Concurrent bisphosphonate or receptor activator of nuclear factor kappa-B (RANK)-ligand directed therapy for prevention of skeletal related events or treatment of osteoporosis is allowed
* Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration; two acceptable methods of birth control thus include the following: condom (barrier method of contraception) AND one of the following is required:

  * Established use of oral, or injected or implanted hormonal method of contraception by the female partner
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner
  * Additional barrier method: occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel film/cream/suppository by the female partner
  * Tubal ligation in the female partner
  * Vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy), for more than 6 months
* Able to swallow the study drug and comply with study requirements
* Estimated life expectancy >= 6 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with prior history of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain arteriovenous malformation or the use of concomitant medications that may lower the seizure threshold or other conditions predisposing to seizure
* Patients who are receiving any other investigational agents
* Patients who are currently taking metformin; prior metformin use is allowed if last dose was 3 months previous to this trial
* Patients with diabetes on a different agent or patients with rheumatoid arthritis taking hydroxychloroquine (Plaquenil)
* Greater than 2 prior therapies in metastatic CRPC (including single-agent docetaxel, abiraterone); abiraterone can only be taken pre-chemotherapy
* Prior cabazitaxel or radium 233 for prostate cancer
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or metformin
* Participation in a previous clinical trial of enzalutamide or an investigational agent that inhibits the androgen receptor (ARN-509) or androgen synthesis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients on antipsychotic medication
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
DLT graded accorded to the National Cancer institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days

SECONDARY OUTCOMES:
Incidence of adverse events graded according to NCI CTCAE version 4.0 | Up to 12 weeks after last dose of study treatment
  The safety analysis population will consist of patients who received any amount of study drug. Clinical and laboratory adverse events will be summarized by coded term and severity. Laboratory values will be plotted over time.
PSA response rate as determined by percent of patients achieving >= 50% PSA decline following initiation of treatment | Up to 12 weeks after last dose of study treatment
  Confidence intervals for the PSA response rate will be calculated using the Clopper-Pearson method, and the PSA response rate will be tested against a null response rate of 50% using an exact binomial test.
PSA progression by Prostate Cancer Working Group (PCWG) 2, defined as the date that a 25% or greater increase and an absolute increase of 2 ng/mL or more from the nadir is documented, which is confirmed by a second value obtained 3 or more weeks later | Up to 12 weeks after last dose of study treatment
  PSA progression by PCWG2 will be assessed and described.
Radiographic disease progression, determined by Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 12 weeks after last dose of study treatment
Progression-free survival | Time from study entry to disease progression in PSA, bone or soft-tissue, symptoms, or death, assessed up to 12 weeks after last dose of study treatment
Time to treatment failure which includes discontinuing therapy because of disease progression, toxicity, or patient withdrawal | Up to 12 weeks after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dall'Era, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States